CLINICAL TRIAL: NCT04794153
Title: Assessing the Muscle Protein Synthetic Response Following the Ingestion of a Variety of Protein Rich Whole Foods Compared to an Isolated Protein Source.
Brief Title: Investigating the Consumption of Different Protein Rich Whole Food Sources on Muscle Growth in Trained Males and Females
Acronym: FFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Marlow Foods Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FFT
Record Dates: First submitted 2021-03-04; First posted 2021-03-11 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Nutritional Intervention Using Protein Rich Whole Food Sources

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Pork (Experimental): Locally sourced
  Interventions: Dietary Supplement: whole food sources
- Salmon (Experimental): Locally sourced
  Interventions: Dietary Supplement: whole food sources
- Mycoprotein (Experimental): Provided by Marlow Foods
  Interventions: Dietary Supplement: whole food sources
- Lentils (Experimental): Red
  Interventions: Dietary Supplement: whole food sources
- Egg (Experimental): Local supplier
  Interventions: Dietary Supplement: whole food sources
- Egg whites (Active Comparator): Local Supplier
  Interventions: Dietary Supplement: whole food sources

INTERVENTIONS:
Dietary Supplement: whole food sources — Foods selected are naturally high in protein and consumed by the general population as part of a meal.

SUMMARY:
Background To date, most of the literature investigating the role of dietary protein in muscle growth has focused on isolated protein sources. However, dietary protein is most commonly consumed within a whole food source. Consuming dietary protein within a whole food matrix may additionally stimulate muscle growth. The idea being, there may be other components within food, capable of producing a greater response.

Objectives: To assess the effect of consuming a variety of whole food sources, on the stimulation of muscle growth compared to an isolated protein source following a single bout of lower body resistance exercise.

Methods Young healthy resistance-trained volunteers will consume a protein rich whole food source, following a bout of lower body resistance exercise. Stable isotope IV infusions and repeated blood and muscle samples will be taken to assess protein digestion and absorption, as well as muscle protein synthesis rates.

Value of Research:

To determine whether whole food sources potentiate muscle protein synthesis rates (and to what extent across whole food sources) compared to an isolated protein source. In doing so, we can further investigate the nutrients involved that may be contributing to this effect.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* BMI 18.5 - 30 kg/m2
* Aged 18 - 40 years
* Structured Resistance training consistently for > 6 months
* A 5-7 day "washout" period from any supplementation

Exclusion Criteria:

* Age >40 years
* Body mass index (BMI) <18.5 or >30 kg/m2
* Any metabolic impairments
* Any cardiovascular impairments
* High blood pressure (≥140/90 mmHg)
* Any gastrointestinal disorders
* Any medications known to affect protein and/or amino acid metabolism
* A personal or family history of epilepsy, seizures or schizophrenia, motor disorder
* Chronic over the counter use of pharmaceuticals (> 1 month)
* Allergic to any of the whole foods included in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Postprandial Muscle protein Synthetic Response following the ingestion of a protein rich whole food source. | 2 years
  84 participants will undergo a single bout of lower body exercise followed by the ingestion of one of the six protein rich whole food sources. Using stable isotope tracer methodology and muscle biopsy samples, the postprandial muscle protein synthetic response will be able to be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Wall, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haigh FAD, Monteyne AJ, Abdelrahman DR, Murton AJ, Finnigan TJA, Theobald HE, Stephens FB, Wall BT. Ingestion of diverse protein-rich whole-foods result in similar post-exercise whole-body and myofibrillar protein synthesis rates compared with a more isolated protein source in young adults. Am J Clin Nutr. 2026 Feb 3:101231. doi: 10.1016/j.ajcnut.2026.101231. Online ahead of print. PMID 41643855